CLINICAL TRIAL: NCT06914011
Title: Multi-center, Randomized, Phase III Trial of Circulating Tumor DNA MRD-Guided Adjuvant Therapy for Curatively Resected Locally Advanced Esophageal Squamous Cell Carcinoma (MRD2START)
Brief Title: Circulating Tumor DNA MRD-Guided Adjuvant Therapy for Curatively Resected Locally Advanced Esophageal Squamous Cell Carcinoma
Acronym: MRD2START
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0183
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adjuvant therapy arm (Experimental): * Participants who underwent upfront surgery without prior neoadjuvant therapy will receive adjuvant chemoradioimmunotherapy in the following sequence:
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for one cycle
    * Concurrent radiotherapy (25 fractions of 1.8 Gy each, with 5 fractions per week) with Tislelizumab 200 mg iv D1, D22, Paclitaxel 50 mg/m2 iv D1, 8, 15, 22, 29, and Carboplatin AUC 2 mg/mL/min D1, 8, 15, 22, 29
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for 1 cycle
    * Tislelizumab D1, in a 6-week cycle for six cycles
  * For participants who underwent neoadjuvant chemoradiotherapy followed by surgery will receive adjuvant chemoimmunotherapy in the following sequence:
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for four cycles
    * Tislelizumab D1, in a 6-week cycle for six cycles
  Interventions: Drug: Tislelizumab
- Follow-up is every 12 weeks for the first 2 years, and then every 24 weeks for up to 5 years. (No Intervention)
- Surveillance arm (No Intervention): •Patients will be followed up without any adjuvant therapy, undergoing CT scans every 12 weeks during the first 2 years after randomization, and thereafter every 24 weeks until 5 years after randomization

INTERVENTIONS:
Drug: Tislelizumab — * Participants who underwent upfront surgery without prior neoadjuvant therapy:
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for one cycle
    * Concurrent radiotherapy (25 fractions of 1.8 Gy each, with 5 fractions per week) with Tislelizumab 200 mg iv D1, D22, Paclitaxel 50 mg/m2 iv D1, 8, 15, 22, 29, and Carboplatin AUC 2 mg/mL/min D1, 8, 15, 22, 29
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for 1 cycle
    * Tislelizumab 400 mg iv D1, in a 6-week cycle for six cycles
  * For participants who underwent neoadjuvant chemoradiotherapy followed by surgery will receive adjuvant chemoimmunotherapy in the following sequence:
    * Tislelizumab 200 mg iv D1, Paclitaxel 175 mg/m2 iv D1, and Carboplatin AUC 5 mg/mL/min iv D1, in a 3-week cycle for four cycles
    * Tislelizumab 400 mg iv D1, in a 6-week cycle for six cycles
  Other Names: Paclitaxel
  Arms: Adjuvant therapy arm

SUMMARY:
This study was a multicenter, randomized, phase 3 trial to determine whether adjuvant chemotherapy including tisleliizumab improves recurrence-free survival compared to follow-up alone without chemotherapy in patients with curatively resected esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
It aims to investigate the efficacy of adjuvant therapy in patients at high risk, as determined by the presence of MRD through cfDNA testing, following curative R0 resection for locally advanced esophageal squamous cell carcinoma.

Patients found to be MRD-positive will be randomly allocated in a 2:1 ratio to either an adjuvant therapy arm or a surveillance arm.

Randomization will be stratified based on the administration of pre-surgery neoadjuvant therapy (yes vs. no), the pathological stage after surgery (0-2 vs. 3-4), and institution.

For participants assigned to the adjuvant therapy arm, those who underwent neoadjuvant chemoradiotherapy followed by surgery will receive adjuvant chemoimmunotherapy comprising paclitaxel + carboplatin + tislelizumab administered every 3 weeks for 4 cycles, followed by tislelizumab monotherapy every 6 weeks for 6 cycles. Patients who had upfront surgery without prior neoadjuvant therapy will receive adjuvant chemoradioimmunotherapy, starting with paclitaxel + carboplatin + tislelizumab every 3 weeks for one cycle, then concurrent radiotherapy (45 Gy in 25 fractions, 1.8 Gy/fraction) with paclitaxel + carboplatin + tislelizumab, followed by an additional cycle of paclitaxel + carboplatin + tislelizumab every three weeks, and concluding with tislelizumab monotherapy every 6 weeks for 6 cycles.

MRD-negative patients are excluded from the phase 3 trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be willing and able to provide written informed consent. 2. Be ≥19 years of age on the day of signing the informed consent form. 3. Have ECOG performance status of 0 or 1 (Appendix 1). 4. Have a histologically confirmed diagnosis of squamous cell carcinoma of the esophagus

  * Patients with tumors of mixed histology (i.e., squamous and non-squamous) are eligible if the predominant histological component is squamous, except when small cell or neuroendocrine elements are present.

    5. Must have completed surgical resection for localized disease, either with prior neoadjuvant chemoradiotherapy or without prior neoadjuvant therapy (i.e., upfront surgery), in accordance with the 8th edition of the AJCC staging system (Appendix 2). Exceptionally, cases with supraclavicular lymph node metastasis as the only M1 lesion are also eligible if the lymph node has been surgically removed.

    6. Must have undergone curative surgery (R0 resection) with negative margins on the resected specimen.

    7. Complete resection must have been performed within 4-16 weeks before randomization.

    8. Must have a documented disease-free status based on a complete physical examination and imaging studies within 4 weeks before randomization. Imaging studies must include CT scans (or MRI) of the chest, abdomen, and pelvis.

    9. Must provide tumor tissue from pre-treatment biopsy (i.e., a biopsy obtained prior to neoadjuvant therapy in cases where neoadjuvant therapy is followed by surgery) or from surgical specimens and baseline blood samples for post-surgery ctDNA-MRD measurement and biomarker analyses.
  * For patients who underwent upfront surgery, surgical tissue is preferred. For those who received neoadjuvant therapy followed by surgery, pre-treatment biopsy tissue is preferred.
  * A FFPE tumor specimen in a paraffin block or 20 (at least 10, with a thickness of 10 µm) freshly cut unstained FFPE slides, along with one H&E-stained slide with tumor-area marking, must be submitted with the associated pathology report. If an insufficient number of slides is available, the decision on patient enrollment can be made in consultation with the Study Sponsor.
  * Peripheral blood of 20 mL must be collected between 3 to 12 weeks after curative surgery for ctDNA testing.

    10. Must be confirmed to have MRD-positive status via postoperative baseline ctDNA testing.

    11. Must have adequate major organ functions as demonstrated by the following laboratory results obtained within 14 days before randomization (these criteria must also be met within 7 days before initiating study treatment in the adjuvant therapy arm):
  * Adequate bone marrow function defined by:
* Absolute neutrophil count (ANC) ≥ 1,500/μL without granulocyte colony-stimulating factor support within 7 days before laboratory testing
* Platelet count ≥ 100 ×103/μL without transfusion within 7 days before laboratory testing • Adequate renal function defined by:
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 50 mL/minute, calculated using the Cockcroft-Gault formula (Appendix 3) or measured by a 24-hour urine collection

  • Adequate hepatic function defined by:
* ALT and AST ≤ 2.5 × ULN
* Total bilirubin ≤ 1.5 × ULN, except for subjects with Gilbert syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who must have a total bilirubin level ≤ 3 × ULN 12. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to randomization. If the urine test is positive or inconclusive, a serum pregnancy test will be required.

  13. Female subjects of childbearing potential randomized to the adjuvant therapy arm must agree to use an adequate method of contraception for the duration of study treatment and for 90 days after the last dose of study treatment.

  14. Non-sterile male subjects randomized to the adjuvant therapy arm with female sexual partner(s) of childbearing potential must agree to use an adequate method of contraception for the duration of study treatment and for 90 days after the last dose of study treatment.

Exclusion Criteria:

* 1. Documented recurrence of esophageal cancer before randomization following curative resection.

  2. Receipt of any treatment aimed at the resected esophageal cancer after curative surgery, including chemotherapy, targeted therapy, immunotherapy, radiotherapy, biologic therapy, investigational agent, or local therapies, except for procedures intended for palliative care (e.g., stent insertion, balloon dilatation, or feeding enterostomy).

  3. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) inhibitor, or any other drug targeting T-cell co-stimulation or checkpoint pathways.

  4. Active autoimmune disease requiring systemic treatment within the 2 years prior to study entry (i.e., using disease-modifying agents, corticosteroids, or immunosuppressive drugs).

  • Replacement therapy (e.g., thyroxine for autoimmune-related hypothyroidism, insulin for type 1 diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.

  5. Condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone or equivalent) or any other form of immunosuppressive therapy within 14 days prior to study entry.

  • Use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids is permitted if there is no active autoimmune disease.
  * A short course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergens) is permitted.

    6. Receipt of a live vaccine within 28 days prior to study entry.
  * COVID-19 vaccines are allowed except for any live vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

    7. Active infection requiring systemic therapy within 14 days prior to study entry.

    8. History of severe hypersensitivity to paclitaxel, carboplatin, or any antibody products.

    9. Known history of, or any evidence of, interstitial lung disease, non-infectious pneumonitis, or pulmonary fibrosis diagnosed based on imaging or clinical findings.
  * Subjects with radiation pneumonitis may be enrolled if radiation pneumonitis is stable (beyond the acute phase) and unlikely to recur.

    10. History of allogeneic stem cell or solid organ transplantation. 11. Malignancies other than esophageal cancer within the 3 years prior to study entry, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%), such as adequately treated non-melanoma skin cancer, superficial bladder cancer, or carcinoma in situ (e.g., cervix, breast, or prostate).
  * Subjects who received endoscopic mucosal resection or dissection for superficial mucosal cancers within the past 3 years are eligible.

    12. Subjects with toxicities attributed to prior anti-cancer therapy, except alopecia, anorexia, fatigue, and hearing loss, that have not resolved to Grade 1 (NCI CTCAE v5.0) or baseline before randomization will be excluded.

    13. Significant cardiovascular impairment within 6 months prior to study entry, including a history of congestive heart failure (New York Heart Association Class III or IV), unstable angina, myocardial infarction, cerebrovascular accident, or cardiac arrhythmia associated with hemodynamic instability.

    14. Any serious or uncontrolled medical disorder that, in the investigator's opinion, may increase the risk associated with study participation or study treatment administration, or compromise the subject's ability to receive protocol therapy.

    15. History or current evidence of any condition, therapy, or laboratory abnormality that could confound trial results, interfere with the subject's participation for the full trial duration, or is not in the best interest of the subject to participate, in the investigator's opinion.

    16. Medical or psychiatric conditions that impair the subject's ability to give informed consent or complete the protocol, or a history of non-compliance.

    17. Known history of Human Immunodeficiency Virus (HIV) infection. 18. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA ≥500 IU/mL (or 2,500 copies/mL), or active hepatitis C virus (HCV) infection:
  * Subjects with chronic hepatitis B (HBV DNA < 500 IU/mL or < 2,500 copies/mL) who are receiving antiviral therapy can be enrolled. Patients with detectable HBsAg or detectable HBV DNA should be managed according to institutional guidelines.
  * Patients with a negative HCV antibody test result at screening or a positive HCV antibody test followed by a negative HCV RNA test result at screening are eligible.

    19. Pregnant or breastfeeding women 20. Any condition requiring treatment with prohibited or restricted concomitant medication or therapy as described in Section 6.2.2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2034-05-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival per RECIST v1.1 | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks

SECONDARY OUTCOMES:
Overall Survival | 5Years
  every visit
Distant metastasis-free survival | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks
Locoregional Recurrence-free survival | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks
Pattern of first recurrence | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks
The incidence and severity of AEs (NCI-CTCAE v5.0) | 5Years
  every visit
Patient-reported outcomes (PROs)-measured HRQoL | 2Years
  * Treatment Period:
    * Adjuvant therapy arm: prior to study treatment on Day 1 of Cycle 1 of the paclitaxel/carboplatin/tislelizumab regimen, prior to dosing at Cycle 1, Cycle 3, and Cycle 5 of tislelizumab monotherapy, and at the EOT/Safety Follow-up visit.
    * Surveillance arm: within 7 days after randomization, and visits at 12W, 24W, 36W, and 48W after randomization
  * Follow-up Period:
  Every 12 weeks during the first two years after randomization
Clearance of ctDNA during and after adjuvant treatment as a predictive biomarker for treatment efficacy, and during surveillance as a prognostic biomarker | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks
ctDNA levels as a predictive biomarker for treatment efficacy and as a prognostic biomarker | 5Years
  Every 12weeks during the first two years after randomization then every 24weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Result] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Result] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338